CLINICAL TRIAL: NCT01621308
Title: Intraperitoneal Insulin Administration as Alternative for Intensive Subcutaneous Insulin Therapy in Patients With Type 1 Diabetes Mellitus.
Brief Title: Intraperitoneal vs Subcutaneous Insulin Administration in Type 1 Diabetes Mellitus
Acronym: IPvsSC
Status: Completed | Type: Observational
Sponsor: Medical Research Foundation, The Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: IPvsSC; NCT01623999 (obsolete NCT alias)
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus type 1; Intraperitoneal insulin administration; Subcutaneous insulin administration; Continuous intraperitoneal insulin infusion
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IP insulin: Patients treated with continuous intraperitoneal insulin infusion using a implantable pump
  Interventions: Other: Mode of insulin administration
- SC insulin: Patients treated with subcutaneous insulin, both multiple daily injections and continuous subcutaneous insulin infusion
  Interventions: Other: Mode of insulin administration

INTERVENTIONS:
Other: Mode of insulin administration — There are no interventions in this observational study. Both treatment groups continue the mode of therapy the patient had before the start of the present study: continuous intraperitoneal insulin infusion with an implantable pump (MIP2007D) or subcutaneous insulin administration with multiple daily injections or continuous subcutaneous insulin infusion.

SUMMARY:
Almost all patients with type 1 diabetes mellitus (T1DM) need insulin treatment permanently. For selected patients who are unable to achieve glycaemic targets with subcutaneous (SC) insulin treatment, continuous intraperitoneal (IP) insulin infusion is an third-line alternative.

Previous studies demonstrate that continuous intraperitoneal insulin infusion (CIPII) using an implantable pump device improves glycaemic control and quality of life in patients with 'brittle' T1DM. Nevertheless, literature comparing IP and SC insulin treatment is scarce.

The primary objective of this study is to compare the effects of IP insulin delivery to SC insulin delivery.The null hypothesis (H0) of the current study holds inferiority of CIPII compared to SC insulin regarding long-term glycaemic control. The alternative hypothesis (H1) is the inverse: CIPII is non-inferior to SC insulin. In summary, H0: CIPII is inferior to the SC insulin treatment H1: CIPII is not inferior to SC insulin treatment

This is an investigator initiated, open label and prospective matched-control study with a non-inferiority design. The trial duration is 36 weeks and is conducted in a single-centre (Isala Clinics, Zwolle). If non-inferiority is established superiority analyses are performed.

ELIGIBILITY:
Case inclusion criteria

* T1DM
* If subjects are on CIPII, they must be included in (8) or
* If subjects are on CIPII, and didn't participate in (8), they must been on CIPII at start of the previous study (8)
* If subjects are on CIPII, they must been on CIPII for the past 4 years without interruptions (>30 days)
* Proper knowledge of the Dutch language.

Case exclusion criteria

* Impaired renal function (plasma creatinine ≥150 µmol/L or glomerular filtration rate as estimated by the Cockcroft-Gault formula ≤50ml/min)
* Cardiac problems (unstable angina or myocardial infarction within the previous 12 months or New York Heart Association class III or IV congestive heart failure
* Mentally handicapped
* Current or past psychiatric treatment for schizophrenia
* Cognitive or bipolar disorder
* Current use or oral corticosteroids or suffering from a condition which necessitated oral or systemic corticosteroids use more than once in the previous 12 months
* Substance abuse, other than nicotine
* Current gravidity or plans to become pregnant during the trial
* Plans to engage in activities that require going >25 feet below sea level
* Any condition that the investigator and/or coordinating investigator feels would interfere with trial participation or evaluation of results.

4.4 Control inclusion criteria

* T1DM
* SC insulin as mode of insulin administration
* If subjects are on SC insulin, they must been on SC insulin for the past 4 years without interruption (>30 days)
* HbA1c at time of matching must be ≥7.0% (53mmol/mol)
* Proper knowledge of the Dutch language.

Control exclusion criteria

* Impaired renal function (plasma creatinine ≥150 µmol/L or glomerular filtration rate as estimated by the Cockcroft-Gault formula ≤50ml/min)
* Cardiac problems (unstable angina or myocardial infarction within the previous 12 months or New York Heart Association class III or IV congestive heart failure
* Mentally handicapped
* Current or past psychiatric treatment for schizophrenia
* Cognitive or bipolar disorder
* Current use or oral corticosteroids or suffering from a condition which necessitated oral or systemic corticosteroids use more than once in the previous 12 months
* Substance abuse, other than nicotine
* Current gravidity or plans to become pregnant during the trial
* Plans to engage in activities that require going >25 feet below sea level
* Any condition that the investigator and/or coordinating investigator feels would interfere with trial participation or evaluation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample consists of the subjects on CIPII, who participated in the crossover study performed by Logtenberg et al. (Diabetes Care 32:1372-1377, 2009) or subjects who already used CIPII at that moment (so, for a minimum of 4 years), and matched controls on SC insulin treatment .
  The inclusion and exclusion criteria of the previous study are described in detail in (Diabetes Care 32:1372-1377, 2009). In brief, it consisted of patients with T1DM, low fasting c-peptide concentrations (<0.20 nmol/L), aged 18 to 70 years, treated with MDI or CSII and intermediate or poor glycaemic control; defined as glycated haemoglobin (HbA1c) ≥7.5% (58 mmol/mol) and/or ≥5 incidents of hypoglycaemia (< 4.0mmol/L) per week.
  If subjects are on SC insulin, they must be able to 'function' as matched control for CIPII patients. The matching procedure, based on age and gender, will take place after patients are being included in the current study.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
glycaemic regulation | 6 months
  HbA1c (mmol/mol)

SECONDARY OUTCOMES:
Percentage time spent in hypo/hyper- and euglycaemia during a 3-7 day 24-hour blood glucose profile using a continuous glucose measurement system (CGMS). | 6 months
Hypoglycaemic episodes | 6 months
Concentrations of IGF-1 and IGFBP | 6 months
Total daily insulin dose. | 6 months
Lipid spectrum | 6 months
Health related quality of life | 6 months
Diabetes related quality of life | 6 months
Diabetes related distress | 6 months
Diabetes related self care | 6 months
Treatment satisfaction | 6 months
body mass index | 6 months
Blood pressure | 6 months
Microvascular complications of diabetes | 6 months
Macrovascular complications of diabetes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Henk JG Bilo, MD PhD FRCP, Study Chair — Isala clinics, Diabetes centre; Peter R Dijk, M.D., Principal Investigator — Isala clinics, Diabetes centre; N Kleefstra, M.D. PhD, Principal Investigator — Isala clinics, Diabetes centre; S JJ Logtenberg, MD PhD, Principal Investigator — Isala clinics, Diabetes centre; University Medical Centre Groningen dept. of internal medicine; Klaas H Groenier, PhD, Principal Investigator — Isala clinics, Diabetes centre; University Medical Centre Groningen dept. of primary medicine
Locations (2):
- Netherlands (2):
  - Diaconessenhuis Hospital, Meppel, Drenthe
  - Isala clinics, Zwolle, Overijssel

REFERENCES:
- [Background] Logtenberg SJ, Kleefstra N, Houweling ST, Groenier KH, Gans RO, van Ballegooie E, Bilo HJ. Improved glycemic control with intraperitoneal versus subcutaneous insulin in type 1 diabetes: a randomized controlled trial. Diabetes Care. 2009 Aug;32(8):1372-7. doi: 10.2337/dc08-2340. Epub 2009 May 8. PMID 19429874
- [Derived] van Dijk PR, Logtenberg SJ, Chisalita SI, Hedman CA, Groenier KH, Gans RO, Kleefstra N, Arnqvist HJ, Bilo HJ. Different Effects of Intraperitoneal and Subcutaneous Insulin Administration on the GH-IGF-1 Axis in Type 1 Diabetes. J Clin Endocrinol Metab. 2016 Jun;101(6):2493-501. doi: 10.1210/jc.2016-1473. Epub 2016 Apr 26. PMID 27115061
- [Derived] van Dijk PR, Logtenberg SJ, Hendriks SH, Groenier KH, Feenstra J, Pouwer F, Gans RO, Kleefstra N, Bilo HJ. Intraperitoneal versus subcutaneous insulin therapy in the treatment of type 1 diabetes mellitus. Neth J Med. 2015 Nov;73(9):399-409. PMID 26582805